CLINICAL TRIAL: NCT03807895
Title: The Effectiveness of an REBT Intervention Program on the Reduction of Career Decision-making Difficulties in High School Pupils
Brief Title: REBT Intervention Program for Career Decision-making Difficulties in High School Pupils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Viktoria Kulcsar, Grad student, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19.175/24.10.2018
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Career Decision-making Difficulties; Worry; Psychological Distress
Keywords: career indecision; career decision-making difficulties; worry; psychological distress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REBT Career Intervention (Experimental): High-school students in the experiment group attend to eight modules of career intervention with rational emotive behavioral therapy (REBT) techniques. The eight modules aim a different component: Psychoeducation, Information about the self and the world of work, Steps of Decision making, Relationship between cognitive distortions/irrational beliefs and emotions, Cognitive Restructuring, Exposure/behavior activation and problem solving, Planning, Goal Setting.
  Interventions: Behavioral: REBT Career Intervention
- Regular Career Intervention (Active Comparator): High-school students in the treatment as usual group attend to eight modules of career intervention with regular career intervention techniques. The eight modules aim a different component: Psychoeducation, Information about the self and the world of work, Steps of Decision making, Problem solving, Planning, Goal Setting.
  Interventions: Behavioral: Regular Career Intervention

INTERVENTIONS:
Behavioral: REBT Career Intervention — Eight sessions of regular career intervention with rational emotive behavioral therapy (REBT) methods.
  Arms: REBT Career Intervention
Behavioral: Regular Career Intervention — Eight sessions of regular career intervention.
  Arms: Regular Career Intervention

SUMMARY:
Career decision-making difficulties are frequent problems for adolescents. Regular intervention or prevention programs mainly provide information for the students about themselves, about the world of work, about their interests and preferences etc. Rational emotive behavioral therapy (REBT), a form of Cognitive behavioral therapy (CBT) provides help for adolescents to efficiently cope with emotional problems (e.g., psychological distress) related to the career decision-making process. The present study aims to investigate the efficiency of an REBT career intervention program implemented in a school setting. School settings are appropriate to deliver group intervention for students. Classes from Romanian public high-schools will be randomized in either intervention or treatment as usual groups.

DETAILED DESCRIPTION:
The intervention will be group based, delivered in 8 sessions, over 8 weeks. Each of the eight modules aimed a different component: Psychoeducation, Information about self and world of work, Steps of career decision-making, Problem solving. Additionally, for the REBT groups: Relationship between cognitive distortions/irrational beliefs and emotions, Cognitive restructuring, Exposure/behavioral activation and emotional problem solving, Maintenance of gaining. Homework would be given at every session. REBT intervention programs delivered in school settings represent ecological modalities to target vulnerable groups. Adolescents will complete assessments at four time points: T1 (baseline), T2 (post-intervention), T3 (3 months follow-up) and T4 (6 months follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents will have ages 16 years to 19 years (11th grade at high school).
* Are attending high school.
* Parents will sign the informed consent and adolescents provide informed assent.

Exclusion Criteria:

* Age below 16 or above 19 years.
* No signed informed consent from the parents.
* Uninterpretable answers on the validation items of the CDDQ (items nr. 7 and 12)

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 235 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Career Decision-making Difficulties Questionnaire (CDDQ; Gati, Krausz, & Osipow, 1996) | Change from baseline career decision-making difficulties up to 24 weeks
  Measure of career decision-making difficulties.

SECONDARY OUTCOMES:
Emotional Distress Profile (PDA; Opris & Macavei, 2005) | Change from baseline distress up to 24 weeks
  Measure of positive emotions, negative functional and negative dysfunctional emotions.
Penn State Worry Questionnaire for Children (PSWQ-C; Chorpita et al., 1997) | Change from baseline worry up to 24 weeks
  Measure of worry for children and adolescents.
General Attitudes and Beliefs Scale Short Form (GABS-SF; Lindner et al., 1999) | Change from baseline irrational beliefs up to 24 weeks
  Measure of Irrational Beliefs.
Beck Depression Inventory for Youth (BDI-Y; Beck, 2005) | Change from baseline depression, anxiety up to 24 weeks
  Measure of depression of adolescents.
Beck Anxiety Inventory for Youth (BAI-Y; Beck, 2005) | Change from baseline anxiety up to 24 weeks
  Measure of anxiety of adolescents.
Career Decision-making Self-Efficacy Short Form (Betz et al., 1996) | Change from baseline career decision-making self-efficacy up to 24 weeks
  Measure of career decision-making self-efficacy.
Multidimensional Life Satisfaction (Seligson, Huebner, & Valois, 2003) | Change from baseline life satisfaction up to 24 weeks
  Measure of five areas of life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Anca Dobrean, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania